CLINICAL TRIAL: NCT02639845
Title: A Novel Eye Drop Application Monitor to Assess Patient Compliance With a Prescribed Regimen
Brief Title: Eye Drop Application Monitor, Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Alexander Eaton (Industry)
Collaborators: California Retina Consultants (Other); Konowal Vision Center (Unknown); Southwest Florida Eye Care (Unknown)
Responsible Party: Sponsor-Investigator, Alexander Eaton, Managing Partner, Retina Health Center
Organization: Retina Health Center (Industry)
Other Study IDs: EDIT Phase I
Record Dates: First submitted 2015-12-18; First posted 2015-12-28 (Estimated); Last update posted 2015-12-28 (Estimated); Status verified 2015-12

CONDITIONS: Cataracts; Retina Surgery; Glaucoma; Any Condition That Requires Ophthalmic Drops
MeSH Terms: conditions — Cataract; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients Prescribed Eye Drops: Patients who are scheduled to receive prescription eye drops due to complications such as cataract surgery, glaucoma, retina surgery, or eye-related condition.

SUMMARY:
The purpose of this study is to determine if an eye drop video monitoring device can accurately assess (as compared to a patient's own log or a proprietary software) the exact amount and time of eye drop delivery to a patient's eye. It is our belief that the experimental device will help patients to be more compliant by: 1) providing a viewable format so patients can see what is happening when they are applying their drops 2) providing greater accuracy to doctors regarding when and how much medication was used 3) providing greater accuracy to doctors and patients regarding how much medication was actually delivered to a patients eye.

DETAILED DESCRIPTION:
Subjects who agree to participate in this study will sign the informed consent form prior to the initiation of any research related procedures. Subjects will be consented by a study coordinator, their physician, or one of the physicians' staff with a strong knowledge of the purpose and design of the clinical trial. There will be two phases to this study: one phase will take place in the clinic, the other will take place at the subjects home. Each subject will participate in each phase. The at home phase will have two arms: one where the subjects are in phase 2 for 1 week, and one where they are in phase 2 for 4 weeks. It is initially anticipated that the 1 week arm will be enrolled first. As the results of the phase 1 come in and patients and physicians get an idea of the ease of using the system, phase 2 will be enrolled. Consented patients who were prescribed an eye drop medication regimen consisting of 1-5 different eye drop medications daily will be asked to participate in this study. Consent and technician assessment will be done by the subject's normal clinician or their designated clinical technician/trial coordinator, all of whom will have been certified for human clinical trials by the Lee Memorial Health System.

The first phase will take place under the controlled clinic environment, where we will assess the ability of the device and reading center to accurately determine the number and volume of drops that get into the eye and the time at which they are instilled as well as log them in an easy to use directory. Five hundred patients, and their designated caregiver if they are unable to apply the drops themselves, will be equipped with the EDAM, trained to use the device, and asked to dispense 10 drops of saline into their eye while in the clinic and being observed by a trained ophthalmic technician. During the application procedure, patients or their designated caregiver, and the observing clinical technician will be asked to write down how many drops were dispensed and if the drop landed in the eye, outside the eye, or half in and half out. All EDAM devices will be returned to the reading center at the Retina Health Center following each use or at the end of each day, along with the subject and technician questionnaires for further assessment. All data will be removed and cleared from the device by the reading center and stored on their secure servers. EDAMs will then be returned to the clinic where they came from for use on other subjects. Accuracy of the written logs (both patients/caregivers and technicians) will be compared to logs created by a technician at the reading center after viewing the application procedure in slow motion and to the read-outs from the drop assessment software.

For the second phase of the trial, these same 500 patients (and their designated caregivers) will be asked to use the EDAM at home for all drop applications for 7 or 28 consecutive days (50 in each group). Patients will be assigned initially to the one week group for short term evaluation of the device and to confirm the ease of use, and safety. Once each patient has completed 1 week of use without any complications, their physician may assign patients to either the four week group or the one week group (if the one week group, they will be done with the study) at their discretion. At the end of each week, subjects and their designated caregivers will be asked to return the EDAM to their clinic which will provide the device to the reading center based at the Retina Health Center. As in the clinical arm, all data will be removed and cleared from the EDAM devices by the reading center and stored on their secure servers for further assessment. EDAMs will then be returned to the clinic where they came from for use on other subjects. At this time, the subject and/or their designated caregiver will also be asked to complete another study questionnaire which will take 5-10 minutes (see appended questionnaire).

Since this is a pilot and exploratory study, it is desirable to allow flexibility to try and identify issues that may develop in both groups prior to undertaking a longer or larger study. Patients will be asked to use the drops routinely. The goal is to see if the EDAM is easy to use, if it captures the desired data, and to get an idea as to patient compliance in a random group of patients. As mentioned, at the end of each week, the patient (with their designated caregiver if applicable) will return to the clinic so a technician can download the accumulated videos and create a log documenting each drop procedure by noting whether each drop made it fully into the eye, half in, not in at all, or if they were unable to make an accurate assessment even with the video recording. This log will be viewed by the physician. The designated care giver may change between eye drop application procedures, but all care givers who assisted in the eye drop procedures must return with the subject to complete a study questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are scheduled to receive prescription eye drops
* Eye drop(s) must be applied at least once a day.
* Caregivers who apply drops for patients

Exclusion Criteria:

* Children (patients < 18 years old)
* Those unable to self-consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive prescription eye drops, one of which must be applied at least once a day.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-11; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Variation from a Prescribed Ophthalmic Drop Regimen | Up to four weeks of monitoring beginning immediately after eye drops are prescribed
  The Eye Drop Application Monitor will be brought to the reading center based at Retina Health Center (Fort Myers, FL) at the end of each use. A trained technician will then document the time of drop delivery and how many drops got in the eye.

CONTACTS AND LOCATIONS:
Overall Officials: Soratree Charoenthongtrakul, Ph.D., Study Director — Retina Health Center
Locations (1):
- Retina Health Center, Fort Myers, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Eaton AM, Gordon GM, Konowal A, Allen A, Allen M, Sgarlata A, Gao G, Wafapoor H, Avery RL. A novel eye drop application monitor to assess patient compliance with a prescribed regimen: a pilot study. Eye (Lond). 2015 Oct;29(10):1383-91. doi: 10.1038/eye.2015.155. Epub 2015 Sep 11. PMID 26358235